CLINICAL TRIAL: NCT02303288
Title: Post-Market Study of the Argus® II Retinal Prosthesis System - France
Status: Completed | Type: Observational
Sponsor: Second Sight Medical Products (Industry)
Responsible Party: Sponsor
Other Study IDs: PM-03-01
Record Dates: First submitted 2014-11-13; First posted 2014-11-27 (Estimated); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Argus II Retinal Prosthesis System — The Argus II System is designed to provide visual function to individuals with severe to profound vision loss due to outer retinal degeneration. It consists of implanted and external components. The implant is an epiretinal prosthesis that is surgically implanted in and around the eye. The external equipment includes glasses and a video processing unit (VPU). The glasses include a miniature video camera, which captures video images, and a coil that sends data and stimulation commands to the implant. The VPU converts the video images into stimulation commands and is body-worn. The Argus II System operates by converting video images into electrical energy that activates retinal cells, delivering the signal through the optic nerve to the brain where it is perceived as light.

SUMMARY:
This is a post-market study of the Argus II Retinal Prosthesis System. The study is being conducted in France. The objective of the study is to obtain data to further demonstrate the effectiveness and evaluate the safety of Argus II System in patients with retinitis pigmentosa who have a bare light perception or worse in both eyes.

DETAILED DESCRIPTION:
This study is a controlled, prospective, multi-centre, single-arm post-market study. All data collected will be obtained from procedures that are performed as part of routine patient case and from non-interventional questionnaires.

Control will consist of three different matched comparisons:

* Post vs. pre-implantation (Baseline) data.
* Prospective within-subject comparisons (implanted vs. non implanted eye)
* Prospective subjects' visual performance Argus II System ON vs Argus II System OFF.

Subjects participating in the study will undergo a Baseline Visit. The Baseline Visit is performed to screen the subject for eligibility for the device and to collect the study baseline assessments. Assessments include a complete eye examination and medical evaluation, retinal photography and Optical Coherence Tomography, Ultrasound A- and B-scans, the photographic flash test, visual acuity tests, the FLORA and a psychosocial evaluation in order to ensure that the subject has realistic expectations about the system. The NEI-VFQ-25 questionnaire will also be administered.

Subjects who are enrolled in the study will undergo a surgery to have the Argus II device implanted. Following implantation surgery, subjects will return to the clinic for periodic clinical follow-up and device fitting. They will also receive training and visual rehabilitation.

Clinical follow-up visits will take place 1 and 2 weeks, 1, 3, 6, 12 and 24 months post-implant. Examinations and tests will be performed as at baseline. In addition, a patient satisfaction, Ease of Use, and Utilization of the System Questionnaire will be administered. Most of the visual function tests and measures will be conducted in both the implanted and fellow eye to provide data on the natural course of the participants' vision loss and as a control for measurements of visual function. In addition, the visual function tests and the FLORA will be done for the implanted eye with the device ON as well as OFF.

Device Fitting refers to the procedure for customizing the Video Processing Unit (VPU) for use by the subject. Device Fitting is typically begins one week post-implant and is completed in approximately 4 sessions.

Beginning approximately one month post-implant, subjects will receive training on how to use the Argus II System. There are two phases of training: system training and visual rehabilitation. During system training, subjects learn basic skills: how to connect the glasses to the VPU, change battery etc., how to control eye movements and RF link, how to scan the environment with head movements and how to use different filters and switch between program settings. During visual rehabilitation, subjects learn how to integrate the use of the Argus II System into their everyday life. Visual rehabilitation sessions will be provided by certified low-vision therapists and/or orientation and mobility specialists and will take place both at the clinic and the subject's home.

ELIGIBILITY:
Inclusion Criteria:

* Are adults, age 25 years or older;
* Have retinitis pigmentosa with visual acuity of bare light perception or worse in both eyes;
* Have previous history of useful form vision;
* If the subject has no residual light perception, the retina must be able to respond to electrical stimulation;
* The subject is willing to provide written, informed consent to participate in the study.

Exclusion Criteria:

* Ocular diseases or conditions that could prevent Argus II from working (e.g. optic nerve disease, central retinal artery or vein occlusion, history of retinal detachment, trauma, severe strabismus, etc.);
* Ocular structures or conditions that could prevent the successful implantation of the Argus II Implant or adequate healing from surgery (e.g. extremely thin conjunctiva; axial length <20.5 mm or > 26 mm; corneal ulcers; choroidal neovascularization in the area of the intended tack location, etc.);
* Ocular diseases or conditions (other than cataracts) that prevent adequate visualization of the inner structures of the eye (e.g. corneal opacity);
* Pre-disposition to eye rubbing;
* Any disease or condition that prevents understanding or communication of informed consent, study demands, and testing protocols, including:

  * cognitive decline including diagnosed forms of dementia and/or progressive neurologic disease,
  * psychiatric disease including diagnosed forms of depression;
  * does not speak a principal language associated with the region, and
  * deafness or selective frequency hearing loss that prevents hearing device alarms and alerts;
* Pregnant or wish to become pregnant during the course of the study;
* Participating in another investigational drug or device study that may conflict with the objectives, follow-up or testing of this study;
* Conditions likely to limit life to less than 1 year from the time of inclusion;
* At the time of the Baseline Visit, suffering from non-ophthalmic serious adverse events (e.g. coma, myocardial infarction, etc.).

Ocular diseases or conditions that could prevent Argus II from working (e.g. optic nerve disease, central retinal artery or vein occlusion, history of retinal detachment, trauma, severe strabismus, etc.);

* Ocular structures or conditions that could prevent the successful implantation of the Argus II Implant or adequate healing from surgery (e.g. extremely thin conjunctiva; axial length <20.5 mm or > 26 mm; corneal ulcers; choroidal neovascularization in the area of the intended tack location, etc.);
* Ocular diseases or conditions (other than cataracts) that prevent adequate visualization of the inner structures of the eye (e.g. corneal opacity);
* Pre-disposition to eye rubbing;
* Any disease or condition that prevents understanding or communication of informed consent, study demands, and testing protocols, including:

  * cognitive decline including diagnosed forms of dementia and/or progressive neurologic disease,
  * psychiatric disease including diagnosed forms of depression;
  * does not speak a principal language associated with the region, and
  * deafness or selective frequency hearing loss that prevents hearing device alarms and alerts;
* Pregnant or wish to become pregnant during the course of the study;
* Participating in another investigational drug or device study that may conflict with the objectives, follow-up or testing of this study;
* Conditions likely to limit life to less than 1 year from the time of inclusion;
* At the time of the Baseline Visit, suffering from non-ophthalmic serious adverse events (e.g. coma, myocardial infarction, etc.).

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with retinitis pigmentosa who have bare light perception or worse in both eyes
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-11-20 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Functional Vision - FLORA | 2 Years
  The impact of the Argus II on subjects' lives (in terms of functional vision and quality of life) as measured by the Functional Low-vision Observer Rated Assessment (FLORA)
Adverse events | 2 Years
  Incidence of procedure- and device-related adverse events

SECONDARY OUTCOMES:
Patient Satisfaction and ease of use of the System | 2 years
  A questionnaire will be administered to track how satisfied or dissatisfied subjects are with the Argus II System, how frequently they use the system, how easy or difficult they think the system is to use, and the ways in which they use the System outside the clinic.
Visual Function | 2 years
  Visual function will be assessed using the following tests:
  * Square Localization: This test assesses subject's light projection.
  * Direction of Motion: This test indicates a subject's ability to detect the direction of a moving object.
  * Grating Visual Acuity: This test is designed to determine a subject's visual acuity using the principles of acuity charts such as ETDRS, modified for extremely low vision. It measures visual acuity between 1.6 to 2.9 logMAR.
  Subjects' performance on the 3 tests above will be compared:
  o Pre-vs. post-implant and. With the Argus II System ON vs. OFF
Functional Vision | 2 years
  The National Eye Institute Visual Function Questionnaire (VFQ-25) will be administered to obtain subjects' self-reported assessment of their vision and what tasks they can perform with their vision (i.e. vision-targeted health status).
Explantation rate | 2 years
  Measure device reliability through explantation rates

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Olivier Barale, MD, Principal Investigator — CHNO des Quinze-Vingts
Locations (3):
- France (3):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris
  - Hôpitaux Universitaires de Strasbourg, Strasbourg